CLINICAL TRIAL: NCT07006272
Title: Cohort Study to Refine the Positioning of Closed-loop Therapy Versus Islet Transplantation in the Management of Patients With Unstable Type 1 Diabetes
Acronym: STABILOOP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC24.0169
Record Dates: First submitted 2025-05-13; First posted 2025-06-05 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: islet transplantation; closed loop
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Closed Loop: Patients who choose te be treated by Closed-Loop in routine care
- Islet Graft: Patients who choose te be treated by Islet Graft in routine care

SUMMARY:
Prospective, multicenter, descriptive cohort (RIPH3 study under the Jardé Act), STABILOOP study aims to describe whether BF may be an appropriate therapeutic option for the cohort of patients who are theoretically candidates for Islet transplantation, by describing Closed-Loop failures at 12 months in patients referred to an expert center for management of unstable diabetes.

ELIGIBILITY:
Inclusion Criteria:

Type 1 diabetic patients describing:

* Significant glycaemic variability defined by the presence of one of these 3 criteria: - Standard deviation > 50% of the glycaemic mean or a MAGE index > 60 mg/dL
* Coefficient of glycaemic variation > 36%
* LBGI index > 5 or HYPOSCORE > 800
* This glycaemic variability must be persistent, i.e. persist for more than 12 months despite optimal diabetes management by a multi-professional team. Optimum management involves :
* Monitoring by a team with expertise in insulin pump and glucose sensor technologies
* Training patients in functional insulin therapy, intensive self-monitoring of blood glucose levels, and prevention and management of situations where there is a risk of hypoglycaemia
* Use of pump and glucose sensor therapy, with interruption before hypoglycaemia
* Reinforced multi-professional support and monitoring, possibly combined with support via telemedicine.
* This glycaemic variability must be considered as severe, i.e. causing unpredictable clinical and metabolic events that impair quality of life, such as severe, disabling and frequent hypoglycaemia (at least 2 Severe Hypoglycaemia with assistance from a third party in the last 12 months or at least 1 Severe Hypoglycaemia with life-threatening consequences in the last 12 months (coma, convulsions or trauma)) or ketosis ketoacidosis.

Exclusion Criteria:

* Patients with type 1 diabetes who do not meet the criteria for islet transplantation
* Patients already fitted with a closed loop
* Kidney transplant patients
* Persons covered by articles L1121-5 to L1121-8 of the CSP (corresponding to all protected persons)
* Persons opposed to participation in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged of minimum 18 years with Type 1 unstable diabetes, eligible to both Islet Transplant of Closed Loop treatement.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Describe Closed Loop (CL) failures at 12 months in patients referred to an expert center for management of unstable diabetes. | 12 months
  Proportion of patients on CL who have had in the year following the introduction of CL therapy : at least 2 severe hypoglycaemias (HS) with assistance from a third party or 1 life-threatening HS (coma or convulsion)

SECONDARY OUTCOMES:
Assess quality of glycaemic control in patients treated with Closed Loop (CL) or Islet Graft (IG) | Before CL initiation or quarterly pre-transplant follow-up, then every 3 months during 2 to 4 follow-up years after CL initiation or 1st IG, depending on the date of inclusion in the study.
  Quality of glycaemic control for CL & IG patients :
  - Data sensor (TIR-TBR-TAR > Glycaemic Target 70-140 & 70-180), reported as percentage of time.
Assess the variation of the glycaemia management index in patients treated with Closed Loop (CL) or Islet Graft (IG) | Before CL initiation or quarterly pre-transplant follow-up, then every 3 months during 2 to 4 follow-up years after CL initiation or 1st IG, depending on the date of inclusion in the study.
  Variation of glycaemia management index for CL & IG patients :
  - Data sensor GMI (%)
Assess glucose variability in patients treated with Closed Loop (CL) or Islet Graft (IG) | Before CL initiation or quarterly pre-transplant follow-up, then every 3 months during 2 to 4 follow-up years after CL initiation or 1st IG, depending on the date of inclusion in the study.
  glucose variability for CL & IG patients :
  - MAGE index
Assess glycaemia variability in patients treated with Closed Loop (CL) or Islet Graft (IG) | Before CL initiation or quarterly pre-transplant follow-up, then every 3 months during 2 to 4 follow-up years after CL initiation or 1st IG, depending on the date of inclusion in the study.
  Data sensor Glycaemia variability for CL & IG patients:
  - CV (%)
Assess the level of mean glucose in patients treated with Closed Loop (CL) or Islet Graft (IG) | Before CL initiation or quarterly pre-transplant follow-up, then every 3 months during 2 to 4 follow-up years after CL initiation or 1st IG, depending on the date of inclusion in the study.
  Level of blood glucose for CL & IG patients :
  * Data sensor average daily blood glucose
Assess hypoglycemia awareness in patients treated with Closed Loop (CL) or Islet Graft (IG) | Before CL initiation or quarterly pre-transplant follow-up, then every 3 months for 1 year then every 6 months for 3 years
  Hypoglycemia awareness for CL & IG patients :
  - Clarke score every 3 months for 1 year then every 6 months for 3 years
Assess balance between hypoglycaemia and hyperglycaemia in patients treated with Closed Loop (CL) or Islet Graft (IG) | Before CL initiation or quarterly pre-transplant follow-up, then every 3 months during 2 to 4 follow-up years after CL initiation or 1st IG, depending on the date of inclusion in the study.
  Balance between hypoglycaemia and hyperglycaemia for CL & IG patients :
  - GRI glycaemic risk index
Assess the evolution of insulin requirement in patients treated with Closed Loop (CL) or Islet Graft (IG) | Before CL initiation or quarterly pre-transplant follow-up, then every 3 months during 2 to 4 follow-up years after CL initiation or 1st IG, depending on the date of inclusion in the study.
  Insulin requirement for CL & IG patients :
  - insulin doses (IU/kg/day)
Assess glycaemia stability in patients treated with Closed Loop (CL) or Islet Graft (IG) | Quarterly pre-transplant follow-up, then every 3 months during 2 to 4 follow-up years 1st IG, depending on the date of inclusion in the study.
  Glycaemia stability for CL & IG patients :
  - HbA1c (%)
Assess renal function in patients treated with Closed Loop (CL) or Islet Graft (IG) | Before CL initiation or quarterly pre-transplant follow-up, then every 3 months during 2 to 4 follow-up years after CL initiation or 1st IG, depending on the date of inclusion in the study.
  Quality of renal function for CL & IG patients :
  - Creatininaemia (µmol/L) to estimate the glomerular filtration rate (mL/min/1.73m²)
Assess occurence of sever diabetic related events in patients treated with Closed Loop (CL) or Islet Graft (IG) | Before CL initiation or quarterly pre-transplant follow-up, then every 3 months during 2 to 4 follow-up years after CL initiation or 1st IG, depending on the date of inclusion in the study.
  For CL & IG patients :
  - sever hypoglycaemia (with assistance from a third party) / ketosis or ketoacidosis
Assess the level of endogenous production of insulin in patients treated with Islet Graft (IG) | Before CL initiation or quarterly pre-transplant follow-up, then every 3 months during 2 to 4 follow-up years after CL initiation or 1st IG, depending on the date of inclusion in the study.
  Level of C-peptide for IG patients :
  - Fasting and stimulated C-peptide (nmol/L)
Assess the quality of the Islet Graft (IG) | Before CL initiation or quarterly pre-transplant follow-up, then every 3 months during 2 to 4 follow-up years after CL initiation or 1st IG, depending on the date of inclusion in the study.
  Quality of islet graft in IG patients :
  - Graft function assessed by IGLS 2.0 score
Assess the antidiabetic management in patients treated with Islet Graft (IG) | Quarterly pre-transplant follow-up, then every 3 months during 2 to 4 follow-up years after 1st IG, depending on the date of inclusion in the study.
  Antidiabetic drug used in IG patients :
  - Presence of antidiabetic drugs other than insulin (metformin, SLGT-2 inhibitor, GLP-1 analogues, DPP4 inhibitor, hypoglycaemic sulphonamides, glinides).
Assessing quality of life related to diabetes disease in patients treated with Closed Loop (CL) or Islet Graft (IG) | Before CL/1st IG, and at 6, 12 and 24 months after CL/1st IG.
  Describing quality of life questionnaires :
  DQOL (Diabetes Quality of Life Measure), score (0-100), higher scores = better quality of life
Assessing global quality of life in patients treated with Closed Loop (CL) or Islet Graft (IG) | Before CL/1st IG, and at 6, 12 and 24 months after CL/1st IG.
  Describing quality of life questionnaires :
  EQ-5D-5L (auto assessed health status questionnaire), score (0-1), higher scores = better health status
Assessing diabetes burden (diabetes-related emotional distress) in patients treated with Closed Loop (CL) or Islet Graft (IG) | Before CL/1st IG, and at 6, 12 and 24 months after CL/1st IG.
  Describing the burden of diabetes/questionnaires :
  T1-DDS (type 1 diabetes distress scale), score (28-168), higher scores = worse outcome
Assessing diabetes burden (fear of hypoglycemia) in patients treated with Closed Loop (CL) or Islet Graft (IG) | Before CL/1st IG, and at 6, 12 and 24 months after CL/1st IG.
  Describing the burden of diabetes:
  HFS (hypoglycemia fear score), score (0-132), higher scores = worse outcome
Assessing diabetes burden (impact and severity of fatigue) in patients treated with Closed Loop (CL) or Islet Graft (IG) | Before CL/1st IG, and at 6, 12 and 24 months after CL/1st IG.
  Describing the burden of diabetes/questionnaires :
  FSS (fatigue severity scale), score (9-63), higher scores = worse outcome
Assess overall patient satisfaction of patients treated with Closed Loop (CL) or Islet Graft (IG) | Before CL/1st IG, then at 6, 12, 24 months post-CL or post 1st IG (or just before a change in treatment modality such as failure of CL or IG)
  Describe patients' overall experience of their treatment modality(ies):
  - DTSQ (diabetes treatment satisfaction questionnaire), score (0-36), higher scores = better treatment satisfaction
Assess overall patient satisfaction of patients treated with Closed Loop (CL) | Before CL/1st IG, then at 6, 12, 24 months post-CL or post 1st IG (or just before a change in treatment modality such as failure of CL or IG)
  Describe patients' overall experience of their treatment modality(ies):
  - INSPIRE questionnaire (insulin dosing systems: perceptions, ideas, reflections, and expectations), score (0-80), higher scores = more positive attitudes or greater perceived benefit/support
Evaluate the clinical course of diabetes treated with Closed Loop (CL) Islet Graft (IG). | Throughout the follow-up period (from 2 to 4 years depending on the date of inclusion in the cohort)
  Clinical evolution criteria to be reported (first occurence):
  HS with assistance of a third party, hypoglycaemic comas, convulsions, cardiovascular events (acute coronary syndrome (ACS), stroke, transient ischaemic attack (TIA), amputations, haemorrhage, thrombosis) cancers, ketosis, ketoacidosis, hospitalisations, infections.
  The data collected will be reported according to the CTCAE v6 classification (classification terminology criteria for adverse events).
Identify the factors associated with Closed Loop (CL) treatment failures (hypoglycaemia) | Throughout the follow-up period (from 2 to 4 years depending on the date of inclusion in the cohort)
  Identification if the "initial number of HS with assistance from a third party" prior to BF therapy is associated with the failure of BF therapy
Identify the factors associated with Closed Loop (CL) treatment failures (diabetes-related emotional distress) | Throughout the follow-up period (from 2 to 4 years depending on the date of inclusion in the cohort)
  Identification if the "initial level of depression/anxiety or distress related to type 1 diabetes (T1-DDS questionnaire)" is associated with the failure of BF therapy
Identify the factors associated with Closed Loop (CL) treatment failures (fear of hypoglycemia) | Throughout the follow-up period (from 2 to 4 years depending on the date of inclusion in the cohort)
  Identification if the "initial level of fear of hypoglycaemia (HSF questionnaire)" is associated with the failure of BF therapy
Identify the factors associated with Closed Loop (CL) treatment failures (HbA1c) | Throughout the follow-up period (from 2 to 4 years depending on the date of inclusion in the cohort)
  Identification if the "initial level of HbA1 (%)" si associated with the failure of BF therapy
Identify the factors associated with Closed Loop (CL) treatment failures (TBR) | Throughout the follow-up period (from 2 to 4 years depending on the date of inclusion in the cohort)
  Identification if the "initial level of % time below 70mg/dL" is associated with the failure of BF therapy
Describe the frequency of occurrence of severe hypoglycaemia with third-party assistance | Throughout the follow-up period (from 2 to 4 years depending on the date of inclusion in the cohort)
  Incidence rate of severe hypoglycaemia with assistance of a third party
Assess the medico-economic impact at 2 years of islet transplantation compared with Closed Loop (CL) therapy from the perspective of the French healthcare system. | At 2 years post-equipment or post-transplant
  The cost differential and the incremental cost-utility ratio (ICUR) will be analysed and expressed as the additional cost per healthy life-year gained with islet transplantation compared with CL therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine LABLANCHE, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (7):
- France (7):
  - HCL - Edouard Herriot Hospital, Lyon, Auvergne-Rhône-Alpes
  - Hospices Civils de Lyon - Lyon Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Strasbourg Civil Hospital, Strasbourg, Grand Est
  - Grenoble University Hospital, La Tronche, ISERE
  - Montpellier University Hospital - Lapeyronnie Hospital, Montpellier, Occitanie
  - Toulouse University Hospital - Hôpital Rangueil, Toulouse, Occitanie
  - APH Paris - LARIBOISIERE Hospital, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No